CLINICAL TRIAL: NCT04915560
Title: Etude de faisabilité Portant Sur un Dispositif de Monitoring Physiologique et d'Une Chaine de téléassistance Des Travailleurs isolés au Sein d'Une société de Nettoyage Industriel.
Brief Title: Feasibility of a Physiological Monitoring for Teleassistance to Isolated Workers in Industrial Cleaning
Acronym: TIGER
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The French committee refused the amendment.
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Ortec International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2021-A01390-41
Record Dates: First submitted 2021-05-25; First posted 2021-06-07 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Work-Related Condition

STUDY DESIGN:
Intervention Model Description: Percentage of valid data obtains from a professional performing an industrial cleaning task wearing a connected T-shirt.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ORTEC Employee (Experimental): ORTEC professional employees performing an industrial cleaning task.
  Interventions: Device: Connected T-shirt

INTERVENTIONS:
Device: Connected T-shirt — Ware of a connected T-shirt

SUMMARY:
The purpose of the study is to test the feasibility of the monitoring of physiological parameters during operations of industrial cleaning

DETAILED DESCRIPTION:
A letter about TIGER study is sent to employees eligible to participate. For volunteers, a written consent is signed after complete oral and written explanation of the protocol is signed.

On the day of the industrial cleaning task, the employee wears the connected t-shirt and performs the cleaning. Data are retrieved on a 5 min interval basis. Physiological parameters above or beyond pre-defined limits are transmitted as potential alarms to an operational teleassistance center. A missing data (Invalid recording) are considered alarms.

The number and causes of alarms are determined after the end of the cleaning task.

ELIGIBILITY:
Inclusion Criteria:

* Employee involved in industrial cleaning task of non-ATEX sites (EXplosive ATmosphere)
* Affiliation to the French National healthcare system
* French speaking employee

Exclusion Criteria:

* Contraindication to the measures or procedures provided for in the study (physical characteristics do not allow measurements to be taken, wounds, etc.)
* Pregnancy
* Inability to understand the study goal
* Employee protected by decision of law

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of T-shirt recording | 12 months
  Percentage of valid data from connected T-Shirt. The physiological data is fed back to an integrator and values for respiratory rate (FR), heart rate (HR), temperature (T °) and activity index are calculated over a period of 5 minutes. These values are only calculated if 15% of the raw data can be used over each period of 5 minutes.

SECONDARY OUTCOMES:
Percentage of alarms processed in less than 3 minutes | 12 months
  Number of alarms processed in less than 3 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Samir HENNI, MD, PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- CHU, Angers, France

IPD SHARING:
Plan to Share IPD: No